CLINICAL TRIAL: NCT03451344
Title: A Community-based Addiction Rehabilitation Electronic System to Improve Recovery Outcomes in Patients With Drug Use Disorder: Protocol for a Randomized Controlled Trial
Brief Title: A Electronic System to Improve Recovery Outcomes in Patients With Drug Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Haifeng Jiang, Attending physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HFJiang
Record Dates: First submitted 2018-01-10; First posted 2018-03-01 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Drug Use Disorders; Addiction, Drug
Keywords: Mobile Health; Illicit drug use; Rehabilitation; Community; China
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To minimize the risk of biased results as much as possible, the persons who conduct the urine tests and complete the evaluation of the ASI will be different from those who provides the intervention. But subjects may talk about the CAREs intervention during the assessment so it is not possible to completely 'blind' the evaluators to the intervention group of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated rehabilitation group (Experimental): Participants will receive the standardized community-based rehabilitation and simultaneously receive a 6-month integrated rehabilitation based on the Community-based Addiction Rehabilitation Electronic System.
  Interventions: Other: Integrated rehabilitation group
- Community-based rehabilitation group (Active Comparator): Participants will receive the standardized community-based rehabilitation.
  Interventions: Other: Community-based rehabilitation group

INTERVENTIONS:
Other: Integrated rehabilitation group — Participant in integrated rehabilitation group needs to visit their corresponding social worker and accept illicit drug test every two months. Social worker will help their corresponding client to apply for social benefits accordingly, and provide counseling irregularly if necessary. The integrated rehabilitation group received the standardized community-based rehabilitation described above and simultaneously received a 6-month integrated rehabilitation based on CAREs (Community-based Addiction Rehabilitation Electronic System).CAREs was developed by the department of addiction research in Shanghai Mental Health Center(SMHC), with functions including education, support, psychological intervention and other functions.
  Arms: Integrated rehabilitation group
Other: Community-based rehabilitation group — Participant in community-based rehabilitation group needs to visit their corresponding social worker for six months and accept illicit drug test every two months. Social worker will help their corresponding client to apply for social benefits accordingly, and provide counseling irregularly if necessary.
  Arms: Community-based rehabilitation group

SUMMARY:
Background: Relapse is very common in patients with illicit drug use disorder and contributes to a series of bad consequences that substantially impact patients' physical and social functions. Due to the limited existence of effective addiction treatment, the majority of patients with drug use disorder could not access help when needing. Mobile health (mHealth) offers a potential solution to improving recovery outcome for patients in community.

Objective: This paper is a protocol for a randomized controlled trial (RCT) of a smart phone application called community-based addiction rehabilitation electronic system (CAREs) . This interactive system consists of an APP for clients and a webpage for service providers, with the aim of teaching clients craving and emergency coping skills and helping service providers to improve work efficiency and effectiveness in community.

Methods: A randomized controlled trial(RCT) will be conducted. Sixty drug illicit users who are newly ordered to undergo community rehabilitation will be recruited from the community in Shanghai. Participants will be 1:1 randomly assigned to receive integrated community rehabilitation by using CAREs or only receiving routine community rehabilitation for 6 months. Corresponding anti-drug social workers will provide service and monitor participants' drug use behavior in accordance with the routine work-flow. Outcomes will be assessed at baseline and in the 6th month. The primary study outcome is the performance on illicit drug urine test which will be carried on regularly twice per week during the study period. Secondary study outcomes include days that participants interact with anti-drug social workers, and the decrease rate of addiction-related issues severity index.

ELIGIBILITY:
Inclusion Criteria:

* (1)Illicit drug users who are newly ordered to undergoing community-based rehabilitation will be recruited for the study.
* (2)Candidates are eligible to participated in if they are aged 20 - 50 years
* (3)Candidates are eligible to participated in if they are meeting the DSM-V (Diagnostic and Statistical Manual of Mental Disorders-V) criteria for substance dependence
* (4)Candidates are eligible to participated in if they are willing to comply with the relevant requirements of the study including using the mobile app
* (5)There is no limitation for Gender when recruiting participant.

Exclusion Criteria:

* (1)Illicit drug users who are not newly ordered to undergoing community-based rehabilitation.
* (2)Candidates' age is less than 20 or older than 50
* (3)Candidates does not meet the DSM-V (Diagnostic and Statistical Manual of Mental Disorders-V) criteria for substance dependence
* (4)Candidates are not able to use the mobile app

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Drug urine test | Up to six months
  The results of drug urine tests will be examined in overall percentage of drug positive samples. Overall percentage of drug positive samples= the number of positive urine tests results / the number of total urine tests (Subject who does not submit urine samples on time during the intervention period or refuses to submit samples even if he/she is present at the site will be considered as having a positive urine test result).

SECONDARY OUTCOMES:
Interacting with anti-drug social workers | Up to six months
  Interaction with anti-drug social workers: The days that participants interact with their corresponding social workers will be collected during the study period. Any phone call, SMS, face-to-face meeting, or communication via CAREs will be considered as interaction happening.
The decrease rate of addiction-related issues severity index | Up to six months
  The Chinese translation of the Addiction Severity Index (ASI) that has good reliability and validity in China will be used to assess the severity of addiction at enrollment and 6 months after enrollment. The descent rate will be counted via dividing the minus value between baseline score and 6-month score by baseline score.
Longest duration of sustained abstinence | Up to six months
  Longest duration of sustained abstinence will be measured by drug urine tests and will be reported in weeks(the most consecutive weeks of drug negative samples).

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Jiang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Haifeng Jiang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Free C, Phillips G, Watson L, Galli L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLoS Med. 2013;10(1):e1001363. doi: 10.1371/journal.pmed.1001363. Epub 2013 Jan 15. PMID 23458994
- [Background] Ingersoll K, Dillingham R, Reynolds G, Hettema J, Freeman J, Hosseinbor S, Winstead-Derlega C. Development of a personalized bidirectional text messaging tool for HIV adherence assessment and intervention among substance abusers. J Subst Abuse Treat. 2014 Jan;46(1):66-73. doi: 10.1016/j.jsat.2013.08.002. Epub 2013 Sep 9. PMID 24029625
- [Background] Mason M, Ola B, Zaharakis N, Zhang J. Text messaging interventions for adolescent and young adult substance use: a meta-analysis. Prev Sci. 2015 Feb;16(2):181-8. doi: 10.1007/s11121-014-0498-7. PMID 24930386
- [Background] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- [Result] Leonhard C, Mulvey K, Gastfriend DR, Shwartz M. The Addiction Severity Index: a field study of internal consistency and validity. J Subst Abuse Treat. 2000 Mar;18(2):129-35. doi: 10.1016/s0740-5472(99)00025-2. PMID 10716096
- [Derived] Xu X, Chen S, Chen J, Chen Z, Fu L, Song D, Zhao M, Jiang H. Feasibility and Preliminary Efficacy of a Community-Based Addiction Rehabilitation Electronic System in Substance Use Disorder: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Apr 16;9(4):e21087. doi: 10.2196/21087. PMID 33861211
- [Derived] Wang Z, Chen S, Chen J, Xu C, Chen Z, Zhuang W, Li X, Zhao M, Haifeng J. A Community-Based Addiction Rehabilitation Electronic System to Improve Treatment Outcomes in Drug Abusers: Protocol for a Randomized Controlled Trial. Front Psychiatry. 2018 Nov 6;9:556. doi: 10.3389/fpsyt.2018.00556. eCollection 2018. PMID 30459653
- See also: UNODC. World Drug Report. 2013 [cited 2014 1 January] — http://www.unodc.org/wdr/